CLINICAL TRIAL: NCT03319732
Title: An Open-Label Study to Evaluate the Long-Term Safety of Arbaclofen Extended-Release Tablets in Multiple Sclerosis Patients With Spasticity (Study OS440-3005)
Brief Title: A Study to Evaluate the Long-term Safety of Arbaclofen Extended-Release Tablets for Patients With Spasticity Due to MS
Acronym: OS440-3005
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RVL Pharmaceuticals, Inc. (Industry)
Collaborators: Osmotica Pharmaceutical US LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OS440-3005
Record Dates: First submitted 2017-10-13; First posted 2017-10-24 (Actual); Results first posted 2022-07-15 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-02

CONDITIONS: Multiple Sclerosis; Spasticity, Muscle
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity | interventions — arbaclofen placarbil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AERT 80 mg (Experimental): Arbaclofen extended release tablet, 20 mg
  Interventions: Drug: Arbaclofen

INTERVENTIONS:
Drug: Arbaclofen — Arbaclofen is the active R enantiomer of baclofen.
  Other Names: AERT

SUMMARY:
Spasticity is a common complication in MS and occurs in up to 84% of patients. The main sign of spasticity is resistance to passive limb movement characterized by increased resistance to stretching, clonus, and exaggerated deep reflexes. Osmotica Pharmaceutical is currently developing arbaclofen extended-release tablets (AERT) for the treatment of spasticity in patients with MS.

DETAILED DESCRIPTION:
This is a multicenter, open-label, long-term extension study to evaluate the safety and tolerability of oral AERT in patients with spasticity due to MS. Subjects from the double blind study (Study OS440-3004) may rollover into this open-label extension study, as well as de novo subjects. The maintenance dose will be 80 mg/day or the highest tolerated dose. Once the subject has reached the maintenance dose, they will remain on that dose for approximately 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18 to 65 years of age, inclusive.
2. An established diagnosis per McDonald Criteria (Polman et al 2011) of MS (either relapsing-remitting [RR] or secondary-progressive [SP] course) that manifests a documented history of spasticity for at least 6 months prior to Baseline.
3. Has participated in Study OS440-3004 or is a new US subject (ie, a de novo subject) who fulfills the inclusion/exclusion criteria.
4. Is willing to continue on open-label treatment with AERT as described in this protocol.
5. If receiving disease-modifying medications (eg, interferons approved for MS, glatiramer acetate, natalizumab, fingolimod, or mitoxantrone), there must be no change in dose for at least 3 months prior to Baseline, and the subject must be willing to maintain this treatment dose for the duration of the study. If receiving AMPYRA® (dalfampridine, fampridine, 4 amino pyridine), subject must be at a stable dose for at least 3 months prior to Baseline.
6. Stable regimen for at least 1 month prior to Baseline for all medications and non pharmacological therapies that are intended to alleviate spasticity.

   a. De novo subjects being considered for enrollment and taking medications indicated for the treatment of spasticity (ie, baclofen, benzodiazepines, cannabinoids, carisoprodol, dantrolene, tizanidine, cyclobenzaprine, any neuroleptic, ropinoprole, tolperisone, and clonidine) must wash out from these medications for a minimum of 21 days by Baseline in order to be eligible for study treatment. De novo subjects found not to meet this criterion will be withdrawn from the study and will be considered screen failures.
7. Absence of infections, peripheral vascular disease, painful contractures, advanced arthritis, or other conditions that hinder evaluation of joint movement.
8. Creatinine clearance, as calculated by the glomerular filtration rate (GFR) using the Modification of Diet in Renal Disease Study (MDRD) formula, of >50 mL/minute.
9. Use of a medically highly effective form of birth control (see Section 7.8 of the protocol) during the study and for 3 months thereafter for women of child-bearing potential (including female subjects).
10. Willing to sign the informed consent form (ICF).

Exclusion Criteria:

1. Any concomitant disease or disorder that has symptoms of spasticity or that may influence the subject's level of spasticity.
2. Inability to rate their level of spasticity or distinguish it from other MS symptoms.
3. Use of high dose oral or intravenous methylprednisolone, or equivalent, within 3 months before Baseline.
4. History of allergy to baclofen or any inactive components of the test formulation.
5. Concomitant use of medications that would potentially interfere with the actions of the study medication or outcome variables (Appendix 5).
6. Pregnancy, lactation, or planned pregnancy during the course of the study and for 3 months after the final study visit.
7. Recent history (within past 12 months) of any unstable psychiatric disease (or yes response to questions 1 or 2 on the Columbia Suicide Severity Rating Scale [C SSRS] at baseline), or current signs and symptoms of significant medical disorders such as severe, progressive, or uncontrolled pulmonary, cardiac, gastrointestinal, hepatic, renal, genitourinary, hematological, endocrine, immunologic, or neurological disease.
8. History of epilepsy.
9. Current significant cognitive deficit, severe or untreated anxiety, severe or untreated depression.
10. Subjects with abnormal micturition that requires indwelling or intermittent catheterization or with lower urinary tract symptoms (LUTS) that result in a score >26 in the Baseline Urinary Symptom Profile - USP© (USP) questionnaire (Appendix 6). Subjects who are proficient in self-catheterization may be included in the study at the investigator's discretion.
11. Current malignancy or history of malignancy that has not been in remission for more than 5 years, except effectively treated basal cell skin carcinoma.
12. Subject has clinically significant abnormal laboratory values, in the opinion of the investigator at Baseline (at Visit 6 for rollover subjects).
13. Any other significant disease, disorder, or significant laboratory finding, including clinically significant abnormal laboratory values or ongoing serious adverse events (SAEs) at Visit 6 (Final Visit) of Study OS440-3004, which, in the opinion of the investigator, puts the subject at risk because of participation, influences the result of the study, or affects the subject's ability to participate.
14. Planned elective surgery or other procedures requiring general anesthesia during the course of the study.
15. History of any illicit substance abuse (eg, alcohol, marijuana, cocaine) or prescription for long-acting opioids within the past 12 months (tramadol use will be allowed).
16. Participation in another clinical research study (with the exception of Study OS440-3004) within 1 month of Baseline.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Jacobs, MD, Study Director — Vice President
Locations (1):
- Neuro Pain Medical Center, Fresno, California, United States

REFERENCES:
- [Derived] Okuda DT, Kantor D, Jaros M, deVries T, Hunter S. Arbaclofen extended-release tablets for spasticity in multiple sclerosis: open-label extension study. Brain Commun. 2023 Feb 7;5(1):fcad026. doi: 10.1093/braincomms/fcad026. eCollection 2023. PMID 36861013

RESULTS

PARTICIPANT FLOW:
Groups:
- AERT 80 mg: Arbaclofen extended release tablet, 20 mg (Two 20-mg tablets twice daily for a total of 80 mg daily dose)
Period: Overall Study
Arm/Group | AERT 80 mg
Started | 323
Completed | 218
Not Completed | 105
Not completed — Adverse Event | 40
Not completed — Withdrawal by Subject | 50
Not completed — MS relapse | 10
Not completed — reason not specified | 5

BASELINE CHARACTERISTICS:
Arm/Group | AERT 80 mg
Number analyzed (Participants) | 323
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 323
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190
  Male | 133
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 312
  More than one race | 1
  Unknown or Not Reported | 4
Height [Mean (Standard Deviation); unit: cm] | 169.6 (8.94)
Weight [Mean (Standard Deviation); unit: kg] | 71.67 (15.704)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: "kg/m^2"] | 24.825 (4.7760)
Total Numeric-Transformed Modified Ashworth Scale-Total Limbs (TNmAS-TL) [Mean (Standard Deviation); unit: units on a scale] — Total Numeric-Transformed Modified Ashworth Scale (TNmAS) is a 6-point scale to measure abnormality in tone or the resistance to passive movements. Higher score is worse outcome.
  For each joint, the minimum score is 0; maximum score is 5. The values for each of the 3 main joints are summed for the limb score. The limb with the highest score is the most affected limb (MAL). The highest possible score for a limb is 15. Limb range: 0 to 15.
  To arrive at total limbs (TL) score the values for all 4 limbs are summed; maximum total limb score is 60. TL range: 0 to 60.
  units on a scale | 13.0 (8.06)
Total Numeric-Transformed Modified Ashworth Scale-Most Affected Limb (TNmAS-MAL) [Mean (Standard Deviation); unit: units on a scale] — Total Numeric-Transformed Modified Ashworth Scale (TNmAS) is a 6-point scale to measure abnormality in tone or the resistance to passive movements. Higher score is worse outcome.
  For each joint, the minimum score is 0; maximum score is 5. The values for each of the 3 main joints are summed for the limb score. The limb with the highest score is the most affected limb (MAL). The highest possible score for a limb is 15. Limb range: 0 to 15.
  To arrive at total limbs (TL) score the values for all 4 limbs are summed; maximum total limb score is 60. TL range: 0 to 60.
  units on a scale | 6.3 (3.25)
Expanded Disability Status Scale (EDSS) [Mean (Standard Deviation); unit: units on a scale] — Expanded Disability Status Scaled (EDSS) is a method of quantifying disability in MS and monitoring changes in the level of disability over time. EDSS range from 1 to 10 in 0.5-unit increments that represent higher levels of disability (lower score is better).
  units on a scale | 4.98 (1.29)
Patient Global Impression of Change (PGIC) [Mean (Standard Deviation); unit: units on a scale] — The patient global impression of change (PGIC) is a standard instrument with a 7-point scale which measures change in the subject's overall status where a value of 1 is very much improved, and value of 7 is very much worse. Score range: 1 to 7; lower score is better. (2= much improved; 3= improved, 4 = no change; 5= minimally worse; 6= much worse).
  units on a scale | 3.3 (1.61)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events, Change in Vital Signs, Clinical Laboratory Test Results, 12-lead ECGs, USP Questionnaire, and C-SSRS Results
Description: Safety and tolerability will be assessed by the monitoring of adverse events volunteered, observed, and elicited by general questions in a non-suggestive manner. Changes in vital signs, clinical laboratory test results, 12-lead ECGs, the urinary symptom profile (USP) questionnaire, and the C-SSRS results will also be assessed.
Time Frame: over 1 year
Population: Safety population included all subjects who received at least one dose of study treatment and had at least one-post dose visit.
Measure: Count of Participants; unit: Participants
Groups:
- AERT 80 mg: Arbaclofen extended release tablet, 20 mg (two 20 mg tablets twice a day for a total of 80 mg daily dose)
Arm/Group | AERT 80 mg
Number analyzed (Participants) | 323
Participants | 276

2. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: Patient Global impression of Change (PGIC) is a scale to evaluate the change in activity limitations, symptoms, emotions, and overall quality of life using scores from 1 to 7 with 1 being no change and 7 being a great deal better, and a considerable improvement that has made all the difference. Minimum value is 1 and the maximum value is 7.
Time Frame: week 60
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AERT 80 mg
Number analyzed (Participants) | 323
units on a scale | 2.7 (1.63)

3. Secondary Outcome: Total Numeric-transformed Modified Ashworth Scale Score or the Most Affected Limb (TNmAS-MAL)
Description: The abbreviated scale title is TNmAS. It is considered the primary clinical measure of muscle spasticity in subjects with neurological conditions. It is a useful 6-point rating scale (0 to 5) to measure abnormality in tone or the resistance to passive movements. Minimum value is 0 and maximum value is 5. A higher score means a worse outcome.
Time Frame: week 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AERT 80 mg
Number analyzed (Participants) | 323
units on a scale | 5.6 (3.22)

4. Secondary Outcome: Expanded Disability Status Scale (EDSS)
Description: Expanded Disability Status Scale (EDSS) is a method of quantifying disability in MS and monitoring changes in the level of disability over time. The EDSS scale ranges from 0 to 10 in 0.5-unit increments that represent higher levels of disability. A score of 0 represents a normal neurological exam, and 10 represents death due to MS.
Time Frame: week 60
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AERT 80 mg
Number analyzed (Participants) | 323
units on a scale | 5.01 (1.3)

ADVERSE EVENTS:
Time Frame: 60 weeks
Arm/Group | AERT 80 mg
All-Cause Mortality (participants affected / at risk) | 1/323
Serious Adverse Events (participants affected / at risk) | 21/323
Other Adverse Events (participants affected / at risk) | 278/323
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AERT 80 mg (N=323)
Acute Myocardial Infarction (Cardiac disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Osteomyelitis (Infections and infestations) | 1
Toxicity to various agents (Infections and infestations) | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Multiple Sclerosis relapse (Nervous system disorders) | 7
Paraparesis (Nervous system disorders) | 1
Restless Legs Syndrome (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Atonic Urinary Bladder (Renal and urinary disorders) | 1
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AERT 80 mg (N=323)
Nausea (Gastrointestinal disorders) | 70
Vomiting (Gastrointestinal disorders) | 29
Asthenia (General disorders) | 61
Gait Disturbance (General disorders) | 20
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 77
Dizziness (Nervous system disorders) | 52
Somnolence (Nervous system disorders) | 41
Headache (Nervous system disorders) | 24
Urinary Tract Disorder (Renal and urinary disorders) | 112

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/32/NCT03319732/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/32/NCT03319732/SAP_002.pdf